CLINICAL TRIAL: NCT05740462
Title: Hydroponic Fortification and Dietary App Effect on Vitamin B12 and Iron (Fe) Status - The Harvest Study, A Randomised Double-blinded Study
Brief Title: Hydroponic Fortification and Dietary App Effect on Nutrients Level (Harvest)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: The Harvest Study
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Iron Deficiency (Without Anemia); B12 Deficiency Vitamin
Keywords: Hydroponic; Dietary app; Salad greens; Iron ferritin; Vitamin B12; vegan recipes
MeSH Terms: conditions — Iron Deficiencies; Vitamin B 12 Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dietary app 1 (Experimental): Dietary app recommends high iron or iron-focused recipes
  Interventions: Behavioral: Recipes consumption; Behavioral: Hydroponic unit
- Dietary app 2 (Sham Comparator): Dietary app recommends standard iron recipes
  Interventions: Behavioral: Recipes consumption; Behavioral: Hydroponic unit
- Hydroponic unit 1 (Experimental): Growing vitamin B12 biofortified plants in a hydroponic unit and will be randomised to dietary app 1 or 2
  Interventions: Behavioral: Recipes consumption; Behavioral: Hydroponic unit
- Hydroponic unit 2 (No Intervention): No hydroponic unit be given to participants and will be randomised to dietary app 1 or 2

INTERVENTIONS:
Behavioral: Recipes consumption — Participants will eat two recipes a day for 17 weeks
  Arms: Dietary app 1; Dietary app 2; Hydroponic unit 1
Behavioral: Hydroponic unit — Participants will grow vitamin B12 biofortified plants for 17 weeks and consume (10 grams) of plant material for 11 weeks.
  Arms: Dietary app 1; Dietary app 2; Hydroponic unit 1

SUMMARY:
Veganism and vegetarianism have clear benefits where they have a lower risk of many health issues. However, they also have a higher risk of nutrients and vitamin deficiency such as iron and vitamin B12. Iron can be found in plant-based food but in varying quantities, whereas vitamin B12 is mainly found in red meat, thus vegans and vegetarians can only take this vitamin in supplements such as tablets. In this study, the investigators are testing two interventions, the consumption of recipes with a certain iron amount to increase iron levels, and the consumption of vitamin B12 biofortified plants to increase serum B12 levels in vegan and vegetarian participants.

DETAILED DESCRIPTION:
Iron is present in plant and animal-derived foods but the fractional absorption of iron from plant foods (that is the percent of iron absorbed from a consumed quantity) is often low (approx 10%) compared to iron from animal sources 25%-30%. It is therefore more challenging for vegans and vegetarians to achieve the Reference Nutrient Intake (RNI) for iron (8.7 mg/day for men over 18 and women over 50, 14.8 mg/day for women aged 18-50), and they are likely to absorb less of that iron and therefore are more likely to become iron depleted.

Plants do not synthesise vitamin B12 and unless fortified, plant-derived foods and beverages do not contain any vitamin B12. the RNI for vitamin B12 in the UK is 1.5 µg/day, therefore it is crucial that vegans and vegetarians take B12 supplements if they don't consume B12-fortified foods or find other ways of incorporating this vitamin into their diets.

The HARVEST study is a 17-week randomised, controlled, double-blinded, parallel dietary intervention study conducted at the Quadram Institute Clinical Research Facility (QI CRF), Norwich, UK. Investigators are seeking vegan or vegetarian women (18 to 50 years old) to test two interventions, iron-specific recipes and B12 biofortified plants grown in a kitchen garden. There are a total of 4 visits (1 screening visit, 2 2-hours visits and 1 short visit). Investigators will assess blood samples for serum ferritin, serum B12 and other iron and B12 biomarkers. Investigators will ask the participant to complete lifestyle questionnaires regarding their dietary pattern, fatigue level and satisfaction and impression of the study tools.

ELIGIBILITY:
Inclusion Criteria:

1. Women over 18 years with a regular menstruation cycle (>21 and <40 days).
2. Has followed a vegan or vegetarian diet that does not include the consumption of meat or fish for at least 1 year.
3. Willing to remain on their background diet for the duration of the study.
4. Those who are on a routine regimen of iron and/or vitamin B12 supplements must maintain the same doses 3 month prior to the study and during the duration of the study.
5. Non-anaemic, haemoglobin (Hb) concentration ≥120 g/L.
6. SF >15 µg/L and <60 µg/L [WHO uses the following cut-offs for context: below 15 µg/L indicates iron deficiency, 16-40 µg/L indicates borderline deficiency, and 41 - 150 µg/L is normal].
7. Body Mass Index (BMI) between 18.5 - 40 kg/m2.
8. Live within 40 miles of the Norwich Research Park.
9. Willing to consume plants grown in the hydroponic unit (e.g., spinach, rocket, mizuna) if they agreed to have a unit.
10. Access to a smartphone or online platform a well as access to the internet.

Exclusion Criteria:

1. Those who have known allergies to the hydroponically grown salad greens (spinach, rocket, mizuna).
2. Flexitarian (consumes meat intermittently) vegetarian.
3. Those with menstruation cycle time periods of <21 or >40-days
4. BMI at screening visit < 18.5 kg/m2 (underweight) and > 40 kg/m2 (severely obese).
5. Those diagnosed with or undergoing treatment for anaemia.
6. Currently pregnant, lactating or trying to conceive.
7. High alcohol consumption, consuming more than 2 drinks per day, can elevate the risk for iron overload.
8. Current smoker or has only ceased in the last 6 months.
9. Diagnosed medical conditions that may impact the study outcomes will be considered on an individual basis.
10. Those with an eating disorders, which may impact the study outcome.
11. On, or about to start, a diet programme such as the 5:2 programme (5:2 programme is where an individual would eat normally for five days a week, and fast for two days a week by reducing calorie consumption).
12. Unable to give written or verbal informed consent.
13. Individuals who cannot understand the written instructions/questionnaires.
14. Unwilling to give GP contact details.
15. Participating in another dietary intervention study or has given blood in another research study during the last 3 months.
16. Any person related to or living with any member of the study team.
17. Those who are part of the Line Manager/supervisory structure of the Chief Investigator.
18. Those who have been asked to self-isolate or have been diagnosed with COVID-19 in the last 14 days. However, participants can be rescreened 7 days after the isolation period.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum ferritin after the dietary app intervention | Week: 0, 6/7 and 17
  Comparison of serum ferritin at baseline and after the intervention
Change of serum B12 after the hydroponic unit intervention | Week: 6/7 and 17
  Comparison of serum B12 at baseline and after the intervention

SECONDARY OUTCOMES:
Change in high sensitivity C-reactive protein (hsCRP) with dietary app (high or standard iron) recipe intervention | Week: 0 to 6/7, 6/7 to 17, and 0 to 17
  comparison of hsCRP at baseline and after dietary app intervention
Change in full blood count (FBC) with dietary app (high or standard iron) recipe intervention | Week: 0 to 6/7, 6/7 to 17, and 0 to 17
  comparison of FBC in venous blood sample at baseline and after dietary app intervention
Change in soluble transferrin receptor (sTfR) with dietary app (high or standard iron) recipe intervention | Week: 0 to 6/7, 6/7 to 17, and 0 to 17
  comparison of sTfR in venous blood sample at baseline and after dietary app intervention
Change in alpha 1 acid glycoprotein (AGP) with dietary app (high or standard iron) recipe intervention | Week: 0 and 17
  comparison of AGP in venous blood sample at baseline and after dietary app intervention
Change in holo-transcobalamin (Holo-TC) after the hydroponic unit (biofortification) intervention | Week: 0 and 17
  Measurement of holo-TC in venous blood sample at baseline and after the hydroponic unit intervention
Change in methylmalonic acid (MMA) after the hydroponic unit (biofortification) intervention | Week: 0 and 17
  Measurement of MMA in venous blood sample at baseline and after the hydroponic unit intervention
Change in total plasma homocysteine (tHcy) after the hydroponic unit (biofortification) intervention | Week: 0 and 17
  Measurement of tHcy in venous blood sample at baseline and after the hydroponic unit intervention

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Kroon, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Quadram Institute Bioscience, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: No